CLINICAL TRIAL: NCT00301405
Title: Open-Label Study of Thalidomide for Chronic Prostatitis/Chronic Pelvic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed. Difficult enrollment of patients with prostatitis.
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Celgene Corporation (Industry); Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-149 IND #74,062
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Prostatitis; Pelvic Pain
Keywords: prostatitis; pelvic pain
MeSH Terms: conditions — Pelvic Pain; Prostatitis | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide (Active Comparator): Open Label drug
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Open label drug

SUMMARY:
To determine the efficacy of thalidomide for treatment of the Chronic Pelvic Pain Syndrome (CPPS).

DETAILED DESCRIPTION:
Prostatitis is the most common urologic diagnosis in men under the age of 50 and the third most common diagnosis in older men. In Chronic Prostatitis (CP) or Chronic Pelvic Pain Syndrome (CPPS), men have lower urinary tract symptoms, pelvic pain, sexual dysfunction and decreased quality of life. Little is known about the cause of CP/CPPS and no definitive therapy exists.

Thalidomide is an immunomodulator (a drug that alters the immune system) and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Thalidomide is approved by the Food and Drug Administration (FDA) for a leprosy skin condition, but not for the treatment of CP or CPPS.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged 18 and older.
2. Male subjects with at least 3 months of symptoms of CP/CPPS who are refractory to other therapies
3. Subjects with a minimum score of 15 on the CPSI.
4. Male subjects must give written informed consent.
5. Male subjects must be willing an able to comply with the most recent version of the FDA-mandated S.T.E.P.S.â Program to include:

   * He understands and can reliably carry out all instructions.
   * He is capable of complying with the mandatory contraceptive measures that are appropriate for male patient registration, and patient surveys as described in the S.T.E.P.S.â program.
   * He has received both oral and written warning of the hazards of taking thalidomide and exposing a fetus to the drug
   * He has received both oral and written warning of the risk of possible contraception failure and of the presence of thalidomide in semen. He has been instructed that he must always use a late condom during any sexual contact with a woman of childbearing potential, even if he has undergone a successful vasectomy.
   * He acknowledges in writing his understanding of these warning and of the need to use a latex condom during any sexual contact with women of childbearing potential, even if he has undergone a successful vasectomy.
   * He agrees NOT to be a sperm or blood donor while being treated with thalidomide -

Exclusion Criteria:

1. Subjects who are female.
2. Subjects with a documented positive urine culture (>100,000 CFU/mL) within the past six months
3. Subjects with duration of symptoms less than three months
4. Subjects with active genital infections
5. Subjects with prior urologic surgeries
6. Subjects with known active or prior genitourinary cancers including renal, ureteral, bladder or prostate
7. Subjects having received prior radiation to the abdominal or pelvic area
8. Subjects with known bladder or ureteral calculi
9. Subjects unable to complete a voiding diary
10. Subjects diagnosed with neuropathy
11. Subjects with neutropenia
12. Subjects with a history of deep venous thrombosis, pulmonary embolism, or hypercoagulable state
13. Any patient who is not willing to comply with the most recent version of the FDA-mandated S.T.E.P.Sâ program
14. Subjects with orthostatic hypotension
15. Subjects with known malignancies in the last 2 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Decrease in pain as measured by visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — William Beaumont Hospital Hospital
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States